CLINICAL TRIAL: NCT03417999
Title: Dose Escalation Pharmacokinetic Study of Intranasal Atomized Dexmedetomidine in Pediatric Patients With Congenital Heart Disease
Brief Title: Pharmacokinetic Study of Intranasal Dexmedetomidine in Pediatric Patients With Congenital Heart Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: All subjects who were enrolled completed the study. However, the PI left the institution and the study was terminated before all cohorts were enrolled.
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Kelly Grogan, Attending Physician, Anesthesia and Critical Care Medicine, Principal Investigator, Children's Hospital of Philadelphia
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 17-014084
Record Dates: First submitted 2018-01-08; First posted 2018-01-31 (Actual); Results first posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2023-09

CONDITIONS: Dexmedetomidine; Congenital Heart Disease
Keywords: Intranasal; Pharmacokinetic; Pediatric
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Cohort 1A:
  * Dexmedetomidine 2 μg/kg
  * Under general oral endotracheal anesthesia
  * 7 subjects age >2 yo and ≤ 6 yo
  * 7 subjects age ≥1 mo and ≤2 yo
  Cohort 1B:
  * Dexmedetomidine 2 μg/kg
  * Under sedation with a natural airway
  * 7 subjects age >2 yo and ≤ 6 yo
  * 7 subjects age ≥1 mo and ≤2 yo
  Interventions: Drug: Dexmedetomidine
- Cohort 2 (Experimental): * Dexmedetomidine 4 μg/kg
  * Under general oral endotracheal anesthesia
  * 7 subjects age >2 yo and ≤ 6 yo
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dose-escalation of atomized intranasal dexmedetomidine
  Other Names: Precedex

SUMMARY:
The main objectives of the study are to determine peak plasma drug concentration levels and corresponding time of dexmedetomidine following intranasal administration in children age ≥1 mo to ≤ 6 yr with congenital heart disease undergoing an elective diagnostic or interventional cardiac catheterization procedure.

DETAILED DESCRIPTION:
The high anxiety levels that children may experience during the preoperative period may be associated with negative medical, psychological, and social consequences. To reduce this stress, and to facilitate separation from parents and the induction of anesthesia, children are often given a sedative prior to undergoing a procedure. Dexmedetomidine is a highly selective a2-adrenergic receptor agonist with sedative, anxiolytic, and analgesic properties. While off-label in its use, the administration of dexmedetomidine by the intranasal route has become a popular and effective technique for sedation in children because it is non-invasive, easy to administer, well tolerated, and relatively fast in onset. Despite this, little consistent data have been published on its onset time, duration of action, or optimal dose. The only available pharmacokinetic (PK) data on dexmedetomidine in pediatric patients is in children who were administered IV dexmedetomidine. We are proposing a prospective open-label inter-subject cohort dose-escalation pharmacokinetic study to obtain peak dexmedetomidine drug concentration level in plasma and the corresponding time point following intranasal administration in the pediatric patient with cardiac disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects age ≥1 mo to ≤6 yo.
2. Subjects must have congenital heart disease.
3. American Society of Anesthesiology (ASA) Physical Status 1-3.
4. Subjects scheduled for elective cardiac interventional or diagnostic catheterization anticipated to last ≥ 3hours.
5. Subjects spontaneously ventilating with a natural airway scheduled for elective cardiac interventional or diagnostic catheterization anticipated to last ≥ 2 hours.
6. Subjects must have reliable intravascular access from which to draw blood samples.

Exclusion Criteria:

1. History of allergic reaction or sensitivity to dexmedetomidine.
2. Nasal pathology preventing the administration of drug.
3. Patients that are on maintenance medications that could inhibit or induce the CYP2A6 enzyme.
4. Cardiac conduction abnormalities defined as second or third degree heart block or pacemaker dependence.
5. Bradycardia, defined by age, upon arrival in the preoperative care area.
6. Hepatic dysfunction defined as a history of hepatic dysfunction AND an Alanine Aminotransferase (ALT) value greater than 2 times normal in the 6 months prior to study drug administration.
7. The subject has received dexmedetomidine or clonidine within 1 week of the study date.
8. BMI >30.
9. Patients previously enrolled in this study.
10. Any investigational drug use within 30 days prior to enrollment.
11. Wards will not be eligible.

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly L Grogan, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective open-label inter-subject cohort dose escalation PK and PD study performed at a since center in a pediatric cardiac catheterization laboratory. Study was approved by IRB on 4/23/18 and the FDA initiation date was 11/29/17. Subjects were enrolled from 06/14/18 through 8/23/21. All study related activities were completed on 10/13/21.
Pre-assignment Details: Some of our subjects were scheduled for a cardiac MRI prior to their heart catheterization. If the MRI answered the clinical question, the heart catheterization was not performed and therefore study drug was not administered.
Groups:
- 2 μg/kg; Subjects Age >2 yo and ≤ 6 yo: Cohort 1A:
  * Dexmedetomidine 2 μg/kg, atomized intranasal
  * Under general oral endotracheal anesthesia
  * Subjects age >2 yo and ≤ 6 yo
- 2 ug/kg; Subjects Age ≥1 mo and ≤2 yo: Cohort 1a:
  * Dexmedetomidine 2 μg/kg, atomized intranasal
  * Under general oral endotracheal anesthesia
  * Subjects age ≥1 mo and ≤2 yo
- 4 μg/kg; Subjects Age >2 yo and ≤ 6 yo: Cohort 2
  * Dexmedetomidine 4 μg/kg, atomized intranasal
  * Under general oral endotracheal anesthesia
  * 7 subjects age >2 yo and ≤ 6 yo
Period: Overall Study
Arm/Group | 2 μg/kg; Subjects Age >2 yo and ≤ 6 yo | 2 ug/kg; Subjects Age ≥1 mo and ≤2 yo | 4 μg/kg; Subjects Age >2 yo and ≤ 6 yo
Started | 10 | 5 (Four subjects received 2 μg/kg and the fifth subject received 1.5 μg/kg due to de-escalation of drug dose based on reaching MTD in cohort.) | 13
Evaluable Subjects ("Completed" is defined here as having received study drug. However, subjects were only considered "evaluable" if they had at least 90 minutes of sampling data to ensure that Tmax was achieved.) | 7 | 3 | 6
Completed ("Completed" is defined here as having received study drug. However, subjects were only considered "evaluable" if they had at least 90 minutes of sampling data to ensure that Tmax was achieved. The number of subjects that were "evaluable" are listed as a Milestone.) | 7 | 5 | 9
Not Completed | 3 | 0 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Procedure cancelled; subject did not receive study drug | 2 | 0 | 2
Not completed — Met exclusion criteria after obtaining consent | 0 | 0 | 1
Not completed — Inadequate study staff available to process samples | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 μg/kg; Subjects Age >2 yo and ≤ 6 yo | 2 ug/kg; Subjects Age ≥1 mo and ≤2 yo | 4 μg/kg; Subjects Age >2 yo and ≤ 6 yo | Total
Number analyzed (Participants) | 10 | 5 | 13 | 28
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 44.5 [38 to 73] | 14 [6.5 to 18] | 40 [28.5 to 64.5] | 38.5 [27 to 59.5]
Age, Customized [Count of Participants; unit: Participants]
  >2 yo and ≤ 6 yo | 10 | 0 | 13 | 23
  ≥1 mo and ≤2 yo | 0 | 5 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8 | 16
  Male | 5 | 2 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4 | 8
  Not Hispanic or Latino | 7 | 4 | 9 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 2 | 1 | 3
  Asian | 1 | 0 | 1 | 2
  White or Caucasian | 7 | 1 | 6 | 14
  Pacific Islander | 0 | 0 | 0 | 0
  Other | 1 | 2 | 5 | 8
  Unknown | 0 | 0 | 0 | 0
  More than one race | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 13 | 28
Weight [Median (Inter-Quartile Range); unit: kilograms] | 15.2 [13.7 to 20.7] | 8.8 [6.1 to 10.9] | 16.1 [13.8 to 17.7] | 14.7 [12.6 to 17.7]
Mixing lesion present [Count of Participants; unit: Participants] — Subjects had a variety of cardiac defects, including those with single versus two ventricle physiology. Subjects were defined by whether they had a mixing lesion or not. These are subjects who had a mixing lesion.
  Participants | 5 | 2 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Samples Obtained Per Subject
Description: Following the administration of atomized intranasal dexmedetomidine, serum samples will be drawn at 0, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240 and 300 minutes post drug administration. This is the number of samples obtained per subject.
Time Frame: Up to 5 hours - 0, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, and 300 minutes post drug administration
Population: Population includes all subjects who received study drug. This included evaluable and non-evaluable subjects.
Measure: Median (Inter-Quartile Range); unit: Samples
Arm/Group | 2 μg/kg; Subjects Age >2 yo and ≤ 6 yo | 2 ug/kg; Subjects Age ≥1 mo and ≤2 yo | 4 μg/kg; Subjects Age >2 yo and ≤ 6 yo
Number analyzed (Participants) | 7 | 5 | 9
Samples | 10 [9 to 10] | 9 [7 to 9] | 10 [6.5 to 10]

2. Primary Outcome: Time of Peak Drug Concentration Level of Dexmedetomidine
Description: Following the administration of atomized intranasal dexmedetomidine, serum samples will be drawn at 0, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240 and 300 minutes post drug administration. The time of peak drug concentration will be determined based on this data.
Time Frame: Up to 5 hours - 0, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, and 300 minutes post drug administration
Population: Analysis population includes subjects who received study drug and had at least 90 minutes of sampling time to ensure that Tmax had been achieved. There was one subject in Cohort 1a who had BLQ for all samples obtained for unknown reasons. This subject's data also not be evaluated.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | 2 μg/kg; Subjects Age >2 yo and ≤ 6 yo | 2 ug/kg; Subjects Age ≥1 mo and ≤2 yo | 4 μg/kg; Subjects Age >2 yo and ≤ 6 yo
Number analyzed (Participants) | 7 | 3 | 6
minutes | 91 [44 to 120] | 30 [15 to 31] | 54 [45 to 106]

3. Primary Outcome: Serum Drug Concentration Levels of Dexmedetomidine
Description: Following administration of atomized intranasal dexmedetomidine, serum samples will be obtained at the following times post administrations: 0, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, and 300 minutes. Peak concentration will be determined based on this data.
Time Frame: Up to 5 hours - 0, 10, 15, 20, 30, 45, 60, 90, 120, 180, 240, and 300 minutes post drug administration
Population: Analysis population includes subjects who received study drug and had at least 90 minutes of sampling time to ensure that Cmax had been achieved. There was one subject in Cohort 1a who had BLQ for all samples obtained for unknown reasons. This subject's data could also not be evaluated.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Groups:
- 2 μg/kg; Subjects Age >2 yo and ≤ 6 yo: Cohort 1A:
  * Dexmedetomidine 2 μg/kg
  * Under general oral endotracheal anesthesia
  * 7 subjects age >2 yo and ≤ 6 yo
Arm/Group | 2 μg/kg; Subjects Age >2 yo and ≤ 6 yo | 2 ug/kg; Subjects Age ≥1 mo and ≤2 yo | 4 μg/kg; Subjects Age >2 yo and ≤ 6 yo
Number analyzed (Participants) | 7 | 3 | 6
pg/mL | 413 [311 to 565] | 570 [315 to 679] | 1000 [978 to 1050]

4. Primary Outcome: Dose-limiting Toxicities (DLT) and/or Maximum Plasma Level > 1000 pg/mL
Description: Dose-limiting toxicities (DLT) include bradycardia, hypotension, new intraventricular conduction abnormality or any serious adverse event possibly, probably, or definitely related to intranasal dexmedetomidine administration that occured after the administration of the intranasal dexmedetomidine and through the completion of PK sampling. Bradycardia, hypotension, or new intraventricular conduction abnormalities that occured after the administration of intravenous dexmedetomidine given by the primary anesthesia team as part of usual clinical care were not considered DLTs but were considered an adverse event. Any events that could not be explained by the intervention that the patient was undergoing were assumed to be related to the study drug.
Time Frame: Subjects were monitored for 6 hours after the administration of study drug.
Population: Population includes any subject who received study drug
Measure: Number; unit: Events
Arm/Group | 2 μg/kg; Subjects Age >2 yo and ≤ 6 yo | 2 ug/kg; Subjects Age ≥1 mo and ≤2 yo | 4 μg/kg; Subjects Age >2 yo and ≤ 6 yo
Number analyzed (Participants) | 7 | 5 | 9
Events | 0 | 2 | 3

ADVERSE EVENTS:
Time Frame: All subjects were monitored for 6 hours after the administration of study drug.
Description: Drug Limiting Toxicities (DLT) were defined as bradycardia, hypotension, new intraventricular conduction abnormality or any serious adverse event related to intranasal dexmedetomidine that occurred after the administration of the intranasal drug and through the completion of PK sampling. Bradycardia, hypotension, or new conduction abnormalities that occured after the administration of intravenous dexmedetomidine given by the primary anesthesia team were considered an adverse event but not a DLT.
Arm/Group | 2 μg/kg; Subjects Age >2 yo and ≤ 6 yo | 2 ug/kg; Subjects Age ≥1 mo and ≤2 yo | 4 μg/kg; Subjects Age >2 yo and ≤ 6 yo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5 | 0/9
Other Adverse Events (participants affected / at risk) | 1/7 | 2/5 | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 μg/kg; Subjects Age >2 yo and ≤ 6 yo (N=7) | 2 ug/kg; Subjects Age ≥1 mo and ≤2 yo (N=5) | 4 μg/kg; Subjects Age >2 yo and ≤ 6 yo (N=9)
Bradycardia not requiring intervention (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) — Bradycardia was a defined adverse event. Bradycardia was defined as a HR <80 bpm in subjects < 1 year old and <60 bpm in subjects >1 year old. This was considered a dose limiting toxicity if if occurred after the administration of study drug.
Hypotension not requiring intervention (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Hypotension is an adverse event. Hypotension is defined as decrease in mean arterial pressure greater than 30% from pressure before administration of study drug. Defined as DLT if occurred after administration of study drug with no other etiology.
New Intraventricular conduction delay (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) — An adverse event was defined as the development of an intraventricular delay following the administration of study drug.
Maximum Plasma Concentration (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) — A maximum plasma concentration >1000 pg/dL was considered a dose-limiting adverse event based on prior data which suggested that when concentrations exceeded this value there was an increased incidence of bradycardia and hypotension.

LIMITATIONS AND CAVEATS:
1. Unable to enroll subjects in Cohort 1B to determine if DEX PK is different in patients spontaneously ventilating with a natural airway versus mechanically ventilated via oral endotracheal tube.
2. Unable to sample long enough to determine elimination phase of IN DEX.
3. Small sample size and heterogenous population limit interpretation of results.
4. COVID delayed enrollment and loss of research personnel.
5. PI left institution prior to completion of study and so study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT03417999/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT03417999/ICF_001.pdf